CLINICAL TRIAL: NCT06165627
Title: Comparison of Clinical Performance of Two Monthly Replacement Toric Soft Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CLV201-P003
Record Dates: First submitted 2023-12-04; First posted 2023-12-11 (Actual); Results first posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Ametropia; Astigmatism
Keywords: Contact lenses; Myopia
MeSH Terms: conditions — Refractive Errors; Astigmatism; Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- T30fA, then Biofinity Toric (Other): Lehfilcon A toric contact lenses worn in Period 1, followed by comfilcon A toric contact lenses worn in Period 2, as randomized. The study lenses will be worn bilaterally (in both eyes) during waking hours for at least 12 hours per day during each wear period (30 days [-1/+3] according to randomization assignment). Study lenses will be removed daily for cleaning and disinfection with CLEAR CARE Cleaning & Disinfecting Solution.
  Interventions: Device: Lehfilcon A toric contact lenses; Device: Comfilcon A toric contact lenses; Device: CLEAR CARE
- Biofinity Toric, then T30fA (Other): Comfilcon A toric contact lenses worn in Period 1, with lehfilcon A toric contact lenses worn in Period 2, as randomized. The study lenses will be worn bilaterally (in both eyes) during waking hours for at least 12 hours per day during each wear period (30 days [-1/+3] according to randomization assignment). Study lenses will be removed daily for cleaning and disinfection with CLEAR CARE Cleaning & Disinfecting Solution.
  Interventions: Device: Lehfilcon A toric contact lenses; Device: Comfilcon A toric contact lenses; Device: CLEAR CARE

INTERVENTIONS:
Device: Lehfilcon A toric contact lenses — Commercially available soft contact lenses worn as indicated
  Other Names: TOTAL30™ for Astigmatism; T30fA
Device: Comfilcon A toric contact lenses — Commercially available soft contact lenses) worn as indicated
  Other Names: Biofinity® Toric; Biofinity Toric
Device: CLEAR CARE — Commercially available hydrogen peroxide-based solution for daily cleaning and disinfection of contact lenses used as indicated
  Other Names: CLEAR CARE® Cleaning & Disinfecting Solution

SUMMARY:
The purpose of this study is to assess the clinical performance of TOTAL30 for Astigmatism (T30fA) soft contact lenses with Biofinity Toric soft contact lenses.

DETAILED DESCRIPTION:
Subjects will be expected to attend 5 office visits and will be dispensed study lenses (per randomization sequence) for 30-day duration of bilateral wear with each study lens (approximately 60 days of lens wear). The total duration of the subject's participation in the study will be approximately 74 days.

ELIGIBILITY:
Key Inclusion Criteria:

* Successful wearer of toric soft contact lenses in both eyes for a minimum of 5 days per week and at least 12 hours per day during the past 3 months;
* Best corrected distance visual acuity (as determined by manifest refraction at screening) better than or equal to 0.10 logMAR in each eye;
* Willing and able to wear the study lenses as specified in the protocol;
* Other protocol-specified inclusion criteria may apply.

Key Exclusion Criteria:

* Biomicroscopy findings at screening that are moderate (Grade 3) or higher and/or corneal vascularization that is mild (Grade 2) or higher; presence of corneal infiltrates;
* Monovision and multifocal contact lens wearers;
* Habitual Biofinity Toric soft contact lens wearers, daily disposable contact lens wearers, and Alcon Toric contact lens wearers in the past 3 months prior to consent;
* Wearing habitual contact lenses in extended wear modality (routinely sleeping in lenses for at least 1 night per week) over the last 3 months prior to enrollment;
* Other protocol-specified exclusion criteria may apply.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 67 (Actual)
Dates: Start 2024-01-23 (Actual); Primary Completion 2024-05-12 (Actual); Study Completion 2024-05-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Lead, Vision Care, Study Director — Alcon Research, LLC
Locations (5):
- United States (5):
  - Kurata Eye Care Center, Los Angeles, California
  - Elsa Pao, OD, Oakland, California
  - Pacific Rims Optometry, San Francisco, California
  - Vision Health Institute, Orlando, Florida
  - ProCare Vision Center, Granville, Ohio

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 67 enrolled, 1 participant was discontinued following randomization but prior to exposure to the study lenses. This reporting group includes all participants exposed to any study lenses evaluated in this study (66).
Units Other Than Participants: eyes
Groups:
- T30fA, Then Biofinity Toric: Lehfilcon A toric contact lenses worn in Period 1, followed by comfilcon A toric contact lenses worn in Period 2, as randomized. The study lenses were worn bilaterally (in both eyes) during waking hours for at least 12 hours per day during each wear period (30 days [-1/+3] according to randomization assignment). Study lenses were removed daily for cleaning and disinfection with CLEAR CARE Cleaning & Disinfecting Solution.
- Biofinity Toric, Then T30fA: Comfilcon A toric contact lenses worn in Period 1, with lehfilcon A toric contact lenses worn in Period 2, as randomized. The study lenses were worn bilaterally (in both eyes) during waking hours for at least 12 hours per day during each wear period (30 days [-1/+3] according to randomization assignment). Study lenses were removed daily for cleaning and disinfection with CLEAR CARE Cleaning & Disinfecting Solution.
Period: First Wear Period (Approx. 30 Days)
Arm/Group | T30fA, Then Biofinity Toric | Biofinity Toric, Then T30fA
Started | 34; 68 eyes | 32; 64 eyes
Completed | 34; 68 eyes | 32; 64 eyes
Not Completed | 0; 0 eyes | 0; 0 eyes
Period: Second Wear Period (Approx. 30 Days)
Arm/Group | T30fA, Then Biofinity Toric | Biofinity Toric, Then T30fA
Started | 34; 68 eyes | 32; 64 eyes
Completed | 34; 68 eyes | 32; 64 eyes
Not Completed | 0; 0 eyes | 0; 0 eyes

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: All subjects/eyes exposed to any study lenses evaluated in this study.
Groups:
- Total: Total of all reporting groups
Arm/Group | T30fA, Then Biofinity Toric | Biofinity Toric, Then T30fA | Total
Number analyzed (Participants) | 34 | 32 | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.6 (7.9) | 31.9 (8.2) | 32.3 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 24 | 41
  Male | 17 | 8 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 5 | 9
  Not Hispanic or Latino | 30 | 27 | 57
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 12 | 12 | 24
  Black or African American | 1 | 3 | 4
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 17 | 17 | 34
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Other | 3 | 0 | 3
  Multi-racial | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 34 | 32 | 66

OUTCOME MEASURES:

1. Primary Outcome: Mean Distance Visual Acuity With Study Lenses at Day 30
Description: Visual Acuity (VA) was assessed for each eye individually with study lenses in place while reading letter charts. VA was recorded in logarithm minimum angle of resolution (logMAR). A logMAR value of 0 equates to 20/20 Snellen VA (normal distance eyesight), with lower logMAR values representing better eyesight.
Time Frame: Day 30 of each wear period. A wear period was 30 days [-1/+3 days] according to randomization assignment.
Population: Safety Analysis Set: All subjects/eyes exposed to any study lenses evaluated in this study with non-missing response. Note, One subject in the Biofinity Toric arm lost a lens on the way to the visit. Hence, the assessment was taken on 1 eye only.
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: eyes
Groups:
- T30fA: Lehfilcon A toric contact lenses worn in Period 1 and worn in Period 2, as randomized.
- Biofinity Toric: Comfilcon A toric contact lenses worn in Period 1 and worn in Period 2, as randomized.
Arm/Group | T30fA | Biofinity Toric
Number analyzed (Participants) | 65 | 62
Number analyzed (eyes) | 130 | 123
logMAR | -0.07 (0.06) | -0.06 (0.06)

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected from time of consent to study exit, up to 74 days.
Description: AEs were obtained through solicited and spontaneous comments from subjects and through observations by the investigator. "At Risk" population for ocular AEs is reported in units of eyes; all other populations are reported in units of subjects. This analysis population includes all subjects/eyes exposed to any study lenses evaluated in this study.
Groups:
- Pretreatment: Events reported in this group occurred before exposure to study lenses.
- T30fA Ocular; T30fA Nonocular: Events reported in this group occurred while exposed to lehfilcon A toric contact lenses.
- Biofinity Toric Ocular; Biofinity Toric Nonocular: Events reported in this group occurred while exposed to comfilcon A toric contact lenses.
Arm/Group | Pretreatment | T30fA Ocular | T30fA Nonocular | Biofinity Toric Ocular | Biofinity Toric Nonocular
All-Cause Mortality (participants affected / at risk) | 0/66 | 0/132 | 0/66 | 0/132 | 0/66
Serious Adverse Events (participants affected / at risk) | 0/66 | 0/132 | 0/66 | 0/132 | 0/66
Other Adverse Events (participants affected / at risk) | 0/66 | 0/132 | 0/66 | 0/132 | 0/66

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.

DOCUMENTS (2):
  • Study Protocol (2023-12-15): https://cdn.clinicaltrials.gov/large-docs/27/NCT06165627/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-03): https://cdn.clinicaltrials.gov/large-docs/27/NCT06165627/SAP_001.pdf